CLINICAL TRIAL: NCT01865396
Title: Effect of Early Palliative Care on Quality of Life of Patients With Advanced Cancer: a Randomised Controlled Trial.
Acronym: IPaC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Vrije Universiteit Brussel (Other); Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012/865
Record Dates: First submitted 2013-05-24; First posted 2013-05-30 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Life-limiting Cancer With Prognosis of Approximately 1 Year

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- early palliative care (Experimental): Interventional palliative care, after diagnosis and once a month.
  Interventions: Behavioral: Interventional palliative care
- Standard care (Active Comparator): Patients will receive the standard oncologic care.
  Interventions: Behavioral: Standard oncologic care

INTERVENTIONS:
Behavioral: Interventional palliative care — Palliative support team will meet the patient soon after diagnosis of incurable disease and will meet the patient at least once a month. The patient will also receive the standard oncologic care.
  Arms: early palliative care
Behavioral: Standard oncologic care — Patients will receive standard oncologic care.
  Arms: Standard care

SUMMARY:
The World Health Organization (WHO) defines palliative care as an approach to improve the quality of life of patients and their families facing life-threatening illness, through prevention and relief of pain and of physical, psychosocial and spiritual problems. The WHO stresses that palliative care is applicable early in the course of the illness together with other therapies that are intended to cure or prolong life, such as chemotherapy or radiation therapy. For the benefit of the patient, palliative care is however often given (too) late in the course of the disease of incurably ill patients.

The aim of our study is to measure the effect of interventional palliative care on quality of life, mood and end-of-life care of patients with advanced cancer and their families. These patients have a limited life expectancy and a high symptom burden, this leads us to suggest that these patients may be benefited with palliative care soon after diagnosis of metastatic disease (interventional palliative care).

The research design of this study is a randomized controlled trial with, on the one hand, an intervention group in which patients and their families receive interventional palliative care in combination with standard cancer care and on the other hand a control group in which patients and their families receive only standard oncologic care. Participants in the intervention group will meet the palliative support team shortly after diagnosis. Afterwards, the palliative support will meet them at least once a month. This intervention focuses on topics such illness understanding, symptom management, decision making and coping with the disease. Participants in the control group will only meet with the palliative support team at the patient's own request or after referral by the oncologist or the nursing staff.

ELIGIBILITY:
Inclusion Criteria:

Patients with life-limiting cancer (prognosis of approximately 1 year) are eligible if:

* Patients are within 12 weeks of referral from an other hospital after receiving first line treatment or within 8 to 12 weeks of a new diagnosis (histological and cytological confirmed):

  * Metastatic and advanced pancreatic, stomach, oesophageal and biliary tract adenocarcinoma;
  * Metastatic or advanced NSCLC (stage IIIB or IV) or metastatic SCLC,
  * Malignant pleural mesothelioma
  * Metastatic or advanced head and neck cancer (stage III or IV)
* Patients are within 12 weeks of progression after receiving treatment and have an prognosis of approximately 1 year:

  * Metastatic and locally advanced colorectal cancer, with progression after second line treatment
  * Metastatic or advanced prostate carcinoma, after second line treatment
  * Advanced breast cancer with visceral and/or brain metastasis, with progression on second or third line treatment
  * Metastatic melanoma,
  * Metastatic or advanced kidney cancer,
  * Metastatic or advanced bladder cancer after first line treatment,

An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 and ability to read and respond to questions in Dutch.

Exclusion criteria:

* Patients under 18 years old
* Patients with impaired cognition
* Patients who met the palliative support team more then once or had a consultation within 6 months of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2013-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Quality of life of the patient and his family caregiver at baseline. | at baseline
  This will be measured with validated questionnaires(EORTC-QLQ C30, McGill QoL, SF-36).
Quality of life of the patient and his family caregiver at 12 weeks. | at 12 weeks
  This will be measured with validated questionnaires (EORTC-QLQ C30, McGill QoL, SF-36).
Quality of life of the patient and his family caregiver, 6-weekly after 12 weeks. | 6-weekly after 12 weeks
  This will be measured with validated questionnaires (EORTC-QLQ C30, McGill QoL, SF-36).

SECONDARY OUTCOMES:
Influence of palliative care on mood and illness-understanding of patients and family caregivers at baseline. | at baseline.
  This will be measured with validated questionnaires (HADS, PHQ-9, illness understanding).
Influence of palliative care on mood and illness-understanding of patients and family caregivers at 12 weeks. | at 12 weeks
  This will be measured with validated questionnaires (HADS, PHQ-9, illness understanding).
Influence of palliative care on mood and illness-understanding of patients and family caregivers 6-weekly, after 12 weeks. | 6-weekly, after 12 weeks.
  This will be measured with validated questionnaires (HADS, PHQ-9, illness understanding).
Influence of palliative care on the decision of physicians with regards to end-of-life-care. | after death of patient
  This will be measured with the questionnaire for decisions wuth regards to end-of-life decision making for physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Vanbelle, MD, PhD, Study Director — University Hospital, Ghent; Luc Deliens, PhD, MD, Study Chair — Vrije Universiteit Brussel and Ghent University
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Vanbutsele G, Pardon K, Van Belle S, Surmont V, De Laat M, Colman R, Eecloo K, Cocquyt V, Geboes K, Deliens L. Effect of early and systematic integration of palliative care in patients with advanced cancer: a randomised controlled trial. Lancet Oncol. 2018 Mar;19(3):394-404. doi: 10.1016/S1470-2045(18)30060-3. Epub 2018 Feb 3. PMID 29402701
- [Derived] Vanbutsele G, Van Belle S, De Laat M, Surmont V, Geboes K, Eecloo K, Pardon K, Deliens L. The systematic early integration of palliative care into multidisciplinary oncology care in the hospital setting (IPAC), a randomized controlled trial: the study protocol. BMC Health Serv Res. 2015 Dec 15;15:554. doi: 10.1186/s12913-015-1207-3. PMID 26666301